CLINICAL TRIAL: NCT01557517
Title: A Randomized Double-Blind Pilot Study of Topical Clobetasol 0.05% Oral Rinse for Oral Chronic Graft-Versus-Host-Disease
Brief Title: Clobetasol for Oral Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Najla El Jurdi, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120068; 12-C-0068
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Oral Chronic Graft vs Host Disease
Keywords: cGVHD; Oral cGVHD; Topical; Oral Rinse; Clobetasol; Oral Graft-Versus-Host Disease; GVHD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clobetasol (Experimental): Patients will rinse oral cavity with 10cc of clobetasol 0.05% for 2 minutes 3 times a day.
  Interventions: Drug: Clobetasol Oral Rinse
- Placebo (Placebo Comparator): Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
  Interventions: Drug: Placebo oral rinse

INTERVENTIONS:
Drug: Clobetasol Oral Rinse — Cycle= up to 4 weeks Patients will rinse oral cavity with 10cc of clobetasol 0.05% oral rinse for 2 minutes 3 times a day.
  Arms: Clobetasol
Drug: Placebo oral rinse — Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
  Arms: Placebo

SUMMARY:
Background:

- Oral graft-versus-host disease (GVHD) is a possible complication of bone marrow transplants. It is the result of the donor cells trying to attack the recipients body. Symptoms include dry mouth, sensitivity and pain when tasting certain spices and flavors, and painful swallowing. Steroids are a possible effective treatment for GHVD, but they can cause side effects when given as pills or injections. Steroids given in a cream or rinse form, applied directly to the site of the symptoms, can have fewer side effects. However, their effectiveness as a rinse has not been tested in the mouth. Researchers want to see if a steroid called clobetasol can be used as a mouth rinse to treat oral GHVD.

Objectives:

- To see if a clobetasol rinse is a safe and effective treatment for oral graft-versus-host disease.

Eligibility:

- Individuals at least 12 years of age who have oral GHVD and are not allergic to clobetasol.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. They will also have an oral exam, a mouth tissue biopsy, and other tests before starting the study drug.
* Participants will be separated into two groups. One group will receive clobetasol; the other will have a placebo liquid.
* Participants will rinse their mouths with the study liquid three times a day after meals for 2 weeks.
* After 2 weeks, participants will have another study visit with blood tests and other exams.
* After the study visit, all participants will start to use the clobetasol rinse. Those who originally had clobetasol will use the rinse for another 2 weeks. Those who originally had a placebo will use the rinse for 4 weeks.
* Participants will have a follow-up exam after the end of treatment....

DETAILED DESCRIPTION:
BACKGROUND:

* Chronic Graft versus Host Disease (cGVHD) is a major late complication of allogeneic hematopoietic stem cell transplantation.
* The oral cavity is the second most commonly affected area in cGVHD and is a major cause of morbidity.
* Clobetasol is a high-potency topical corticosteroid widely used for a variety of inflammatory disorders of the skin and oral mucosa.
* Treatment of oral cGVHD by topical agents is an attractive strategy to potentially avoid adverse effects associated with systemic immunosuppression.

OBJECTIVES:

- To investigate efficacy of topical clobetasol 0.05% oral rinse for oral chronic graft versus-host disease (cGVHD)

ELIGIBILITY:

- Patients age 12-99 years with clinically significant oral cGVHD.

DESIGN:

* This is a randomized, double blind, placebo-controlled, pilot study of clobetasol 0.05% topical oral rinse with an open label extension period.
* Patients will rinse oral cavity with 10cc of clobetasol 0.05% or placebo oral rinse for 2 minutes 3 times a day.
* Treatment duration will be for 2 weeks in the randomized phase and 2-4 weeks in the open label phase.
* Up to 40 patients will be enrolled on this pilot trial until 34 evaluable patients are assessed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 12 years 99 years.
* Diagnosis: clinically significant oral chronic graft versus host disease (cGVHD) after allogeneic hematopoietic stem cell transplant (HSCT) with severity score of at least 2 on erythema subset and/or at least 1 on ulceration subset and a composite score greater than or equal to 20 of the Oral Mucositis Rating Scale (OMRS) scale confirmed by the principal investigator (PI), clinical study chair (CSC), or lead associate investigator (LAI).
* Hematologic Function: Patients must have a platelet count greater than or equal to 20,000/microL at the time of the initial evaluation.
* Informed Consent: All patients or their legal representative (for patients <18 years old) must sign an institutional review board (IRB) approved informed consent document (cGVHD natural history protocol 04-C-0281 or any National Cancer Institute (NCI) protocol allowing for screening procedures) prior to performing studies to determine patient eligibility. After confirmation of patient eligibility all patients or their legal representative must sign the protocol specific informed consent. For pediatric patients age appropriate assent will be obtained in accordance with National Institutes of Health (NIH) guidelines.
* Patients must be able to rinse and expectorate study medication rather than swallow it. Female patients must be willing to practice birth control (including abstinence) during and for two months after treatment, if of childbearing potential.
* Patients must have the ability and willingness to come to Clinical Center for bi-weekly follow-up appointments.
* No change in systemic immunosuppressive therapy (type or intensity level) within 2 weeks prior to enrollment.
* A 7-day washout period is required if patients are currently using another oral topical treatment for mouth lesions. Patients currently using clobetasol oral topical treatment are not eligible for this study.

EXCLUSION CRITERIA:

* Documented hypersensitivity to clobetasol.
* Use of clobetasol ointment intra-orally at any time during the last 6-month period.
* Pregnant or breast-feeding females due to possible toxicity to the fetus or infant.
* Inability to understand the investigational nature of the study to provide informed consent.
* Patients who, for medical or other reasons, are unable to comply with the study procedures.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imanguli MM, Pavletic SZ, Guadagnini JP, Brahim JS, Atkinson JC. Chronic graft versus host disease of oral mucosa: review of available therapies. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Feb;101(2):175-83. doi: 10.1016/j.tripleo.2005.08.028. PMID 16448918
- [Background] Pavletic SZ, Lee SJ, Socie G, Vogelsang G. Chronic graft-versus-host disease: implications of the National Institutes of Health consensus development project on criteria for clinical trials. Bone Marrow Transplant. 2006 Nov;38(10):645-51. doi: 10.1038/sj.bmt.1705490. Epub 2006 Sep 18. PMID 16980994
- [Background] Flowers ME, Parker PM, Johnston LJ, Matos AV, Storer B, Bensinger WI, Storb R, Appelbaum FR, Forman SJ, Blume KG, Martin PJ. Comparison of chronic graft-versus-host disease after transplantation of peripheral blood stem cells versus bone marrow in allogeneic recipients: long-term follow-up of a randomized trial. Blood. 2002 Jul 15;100(2):415-9. doi: 10.1182/blood-2002-01-0011. PMID 12091330
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0068.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Clobetasol Followed by Assessment + 2 Weeks Clobetasol: Patients will rinse oral cavity with 10cc of clobetasol 0.05% for 2 minutes 3 times a day.
  Clobetasol Oral Rinse: Cycle= up to 4 weeks Patients will rinse oral cavity with 10cc of clobetasol 0.05% oral rinse for 2 minutes 3 times a day.
- Placebo Followed by Clobetasol: Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
  Placebo oral rinse: Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
Period: Overall Study
Arm/Group | Clobetasol Followed by Assessment + 2 Weeks Clobetasol | Placebo Followed by Clobetasol
Started | 19 | 21
Completed | 17 | 17
Not Completed | 2 | 4
Not completed — Death | 1 | 0
Not completed — Refused further treatment | 0 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Pt declined before treatment started | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobetasol | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.09 (14.52) | 41.4 (16.53) | 42.75 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 13 | 10 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 3 | 6
  White | 15 | 13 | 28
  Asian | 0 | 3 | 3
  Unknown | 1 | 0 | 1
  Multiple Race | 0 | 2 | 2
  Mexican, Puerto Rican, Cuban, Central or So. Amer. | 3 | 3 | 6
  Not meeting definition for Hispanic or Latino | 16 | 18 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response as Assessed by the 273-point Oral Mucositis Rating Scale (OMRS) Who Received Topical Clobetasol 0.05% Oral Rinse for Oral Chronic Graft-versus-host-disease (cGVHD) During a Four-week Treatment Period
Description: Mucosal changes were assessed by the Oral Mucositis Rating Scale. The primary endpoint was evaluated using the OMRS. Oral tissue changes are rated on a scale of 0-3 compared with normal oral tissue (0-normal/no change, 1-mild change, 2-moderate change, and 3-severe change). Total score is the sum of all OMRS items with a possible range of 0. Total score is the sum of all OMRS items with a possible range of 0-273. Lower score=more normal oral mucosa. There is no standard definition of response in this field. Definitions we used in this pilot study to grade the response to study intervention are: Progress of 25% of initial score (rounded to the closest number) on the OMRS scale. Completion (PD) is defined as an increase of 25% of initial score (rounded to the closest number). Partial Response (PR) is defined as a decrease Response (CR) is defined as a PR plus a score of 0 on the erythema and ulceration components. Stable Disease (SD) does not meet criteria for progression or response.
Time Frame: At 4 weeks on active treatment
Population: 18/19 are analyzed in the Clobetasol arm/group because one participant declined participation before treatment started.
Measure: Number; unit: percentage of participants
Groups:
- Clobetasol (2-week): Patients will rinse oral cavity with 10cc of clobetasol 0.05% for 2 minutes 3 times a day.
  Clobetasol Oral Rinse: Cycle= up to 4 weeks Patients will rinse oral cavity with 10cc of clobetasol 0.05% oral rinse for 2 minutes 3 times a day.
- Placebo (2-week): Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
  Placebo oral rinse: Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
- Combined Group 4-week Data: Patients will rinse oral cavity with 10cc of clobetasol 0.05% oral rinse for 2 minutes 3 times a day. This group includes patients initially randomized to the clobetasol group as well as the patients initially randomized to placebo, who crossed over to the clobetasol 0.05% oral rinse group after 2 weeks of placebo use and the interim assessment and then completed 4 weeks of clobetasol rinse use.
Arm/Group | Clobetasol (2-week) | Placebo (2-week) | Combined Group 4-week Data
Number analyzed (Participants) | 18 | 21 | 31
percentage of participants
  Progressive Disease | 0 | 0 | 0
  Partial Response | 72 | 9 | 72
  Complete Response | 0 | 0 | 19
  Stable Disease | 28 | 91 | 9

2. Secondary Outcome: Percent Change in Participants' Raw Score of Oral cGVHD Related Pain on a 0-10 Rating Scale
Description: Oral cavity pain was assessed by an oral cavity specific quality of life questionnaire. Pain was rated based on a 0-10 rating scale on which subjects selected a single integer. 0 = no pain and 10 = worst pain. A negative value indicates an increase in oral pain. A positive value indicates an improvement in patient-perceived oral pain.
Time Frame: Baseline to Day 14 and baseline to Day 28
Population: 18/19 are analyzed in the Clobetasol grp because one participant declined participation before treatment started. Clobetasol and Placebo grps were not assessed separately at Day 28. Only those pts who completed 4 wks of active clobetasol treatment and did not have an active oral infection at the 4 week timepoint were included in the final analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Clobetasol | Placebo | Combined Group 4-week Data
Number analyzed (Participants) | 18 | 21 | 31
Percent change
  Day 14 | 13 (116) | 21 (67) | 31 (86)
  Day 28 | NA (NA) — Day 28 data for this Clobetasol Arm/Group is collapsed within the Combined Group 4-week data Arm/Group. | NA (NA) — Day 28 data for this Placebo Arm/Group is collapsed within the Combined Group 4-week data Arm/Group. | 45 (146)

3. Secondary Outcome: Percent Change in Participants' Raw Score of Oral cGVHD Related Sensitivity on a 0-10 Rating Scale
Description: Oral cavity sensitivity was assessed by an oral cavity specific quality of life questionnaire. Sensitivity was rated based on a 0-10 rating scale on which subjects selected a single integer. 0 = no sensitivity and 10 = worst sensitivity. A negative value indicates an increase in oral sensitivity. A positive value indicates an improvement in patient-perceived oral sensitivity.
Time Frame: Baseline and 4 weeks on active treatment
Population: 18/19 are analyzed in the Clobetasol grp because one participant declined participation before treatment started.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Clobetasol | Placebo | Combined Group 4-week Data
Number analyzed (Participants) | 18 | 21 | 31
Percent change | 39 (168) | 19 (62) | 41 (106)

4. Secondary Outcome: Percent Change in Participants' Raw Score of Oral cGVHD Related Dryness on a 0-10 Rating Scale
Description: Oral cavity dryness was assessed by an oral cavity specific quality of life questionnaire. Dryness was rated based on a 0-10 rating scale on which subjects selected a single integer. 0 = no dryness and 10 = worst dryness. A negative value indicates an increase in patient-perceived oral dryness. A positive value indicates an improvement in patient-perceived oral dryness.
Time Frame: Baseline and 4 weeks on active treatment
Population: 18/19 are analyzed in the Clobetasol grp because one participant declined participation before treatment started.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Clobetasol | Placebo | Combined Group 4-week Data
Number analyzed (Participants) | 18 | 21 | 31
Percent change | 8 (115) | 15 (229) | 30 (111)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Clobetasol During Pharmacokinetic Testing
Description: Steady-state pharmacokinetics of systemic clobetasol were assessed following a single 2 min oral rinse of 0.05% clobetasol on day 14 (1 patient collected on day 12). A noncompartmental pharmacokinetic assessment was performed using WinNonlin v5 (Pharsight Corp, Mountain View, CA) from three sampling times (pre-rinse, 15-45 min post-rinse, and 90-120 min post-rinse). Plasma concentrations of clobetasol were measured using a newly designed and validated LC-MS/MS assay, with a lower limit of quantification of 0.05 ng/mL. The maximum plasma concentrations (CMAX) were recorded as observed values and the area under the plasma-concentration time curve using all three sampling time points (AUCALL) was calculated using the Linear Trapezoidal rule.
Time Frame: pre-rinse, 15-45 min post-rinse, and 90-120 min post-rinse
Population: Per protocol, pharmacokinetic testing was only done on the first 10 patients in the clobetasol group. We are reporting a calculation based on these 3 time points, not a number that can be reported at 3 discrete times.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Clobetasol
Number analyzed (Participants) | 10
ng/mL | 0.818 (0.649)

6. Secondary Outcome: Plasma Concentrations of Clobetasol Mouth Rinse in cGVHD Patients at Baseline (Day 0) and Day 28
Description: Peripheral blood was drawn at baseline and day 28 of clobetasol rinse use, and clobetasol levels were measured in the blood sample. Plasma concentrations of clobetasol were measured using a validated LC-MS/MS assay with a lower limit of quantification of 0.05 ng/mL. Any values below detectable limit or with no peak were adjusted to 0.
Time Frame: Baseline Day 0 and Day 28
Population: 37/40 participants are included in this laboratory assessment as interpretable data was not available for 3 patient samples.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combined Group 4-week Data
Number analyzed (Participants) | 37
ng/mL
  Baseline (Day 0) | 0.0146 (0.0578)
  Day 28 | 0.329 (0.343)

7. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 62 months and 12 days.
Population: 18/19 are analyzed in the Clobetasol arm/group because one participant declined participation before treatment started.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo First (During Clobetasol Phase Only); Placebo (During 2-week Placebo Phase Only): Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
  Placebo oral rinse: Patients will rinse oral cavity with 10cc of placebo oral rinse for 2 minutes 3 times a day.
Arm/Group | Clobetasol | Placebo First (During Clobetasol Phase Only) | Placebo (During 2-week Placebo Phase Only)
Number analyzed (Participants) | 18 | 21 | 21
Participants | 17 | 21 | 6

8. Secondary Outcome: Time to Maximum Plasma Concentration (Cmax) of Clobetasol
Description: as for outcome 5
Time Frame: pre-rinse, 15-45 min post-rinse, and 90-120 min post-rinse
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Clobetasol
Number analyzed (Participants) | 10
hours | 1.27 (0.59)

9. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve for All Time Points
Description: as for outcome 5
Time Frame: pre-rinse, 15-45 min post-rinse, and 90-120 min post-rinse
Population: Per protocol, pharmacokinetics testing was only done on the first 10 patients in the clobetasol group.
Measure: Mean (Standard Deviation); unit: Hr*ng/mL
Arm/Group | Clobetasol
Number analyzed (Participants) | 10
Hr*ng/mL | 0.974 (0.729)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 62 months and 12 days.
Description: 18/19 are participants in the Clobetasol arm/group because one participant declined participation before treatment started.
Arm/Group | Clobetasol | Placebo First (During Clobetasol Phase Only) | Placebo (During 2-week Placebo Phase Only)
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/18 | 4/21 | 0/21
Other Adverse Events (participants affected / at risk) | 16/18 | 21/21 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol (N=18) | Placebo First (During Clobetasol Phase Only) (N=21) | Placebo (During 2-week Placebo Phase Only) (N=21)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — enlarging mediastinal lymphadenopathy
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol (N=18) | Placebo First (During Clobetasol Phase Only) (N=21) | Placebo (During 2-week Placebo Phase Only) (N=21)
Adrenal insufficiency (Endocrine disorders) | 10 (10) | 11 (11) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 8 (8) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 4 (6) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 7 (9) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (12) | 8 (8) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0)
Diarrhea (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — EBV low positive
Insomnia (Psychiatric disorders) | 5 (5) | 7 (7) | 1 (1)
Mucosal infection (Infections and infestations) | 5 (8) | 6 (6) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 3 (3) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicitis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — CMV reactivation
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT01557517/Prot_SAP_001.pdf
  • Informed Consent Form (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT01557517/ICF_002.pdf